CLINICAL TRIAL: NCT03165565
Title: Facilitating Treatment Entry and Family Planning in Substance-using NICU Mothers
Brief Title: Facilitating Treatment Entry and Family Planning in Substance-using Neonatal Intensive Care Unit (NICU) Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Angela L Stotts, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0990; R34DA041465 (NIH)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI and ACT (Experimental): Participants will receive behavioral therapy including Motivational Interviewing (MI) and Acceptance and Commitment Therapy (ACT).
  Interventions: Behavioral: Motivational Interviewing (MI) and Acceptance and Commitment Therapy (ACT)
- Conventional Care (Active Comparator): Conventional care from the hospital for NICU mothers who test positive for drug use, which includes visits and resources from hospital social workers.
  Interventions: Behavioral: Conventional Care

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) and Acceptance and Commitment Therapy (ACT) — Participants will receive Motivational Interviewing (MI) and Acceptance and Commitment Therapy (ACT).
  Arms: MI and ACT
Behavioral: Conventional Care — Conventional care from the hospital for NICU mothers who test positive for drug use, which includes visits and resources from hospital social workers.
  Arms: Conventional Care

SUMMARY:
The purpose of this pilot study is to assess whether the hospital-based, adaptive behavioral intervention strategy promotes treatment entry and reduces risk of additional substance-exposed pregnancies (SEPs), as well as HIV and Hepatitis C Virus (HCV) risks among substance-using NICU mothers. Additionally, to assess whether the intervention increases use of professional obstetrical/gynecological resources for contraception to reduce substance-exposed pregnancies (SEPs).

ELIGIBILITY:
Inclusion Criteria:

* have an infant in the NICU at Children's Memorial Hermann Hospital (CMHH)
* have a positive urine drug screen at delivery or have an infant with a positive urine or meconium drug screen or self-reported drug use to a healthcare provider or had a documented positive drug screen during pregnancy
* have access to a telephone.

Exclusion Criteria:

* currently attending substance abuse treatment
* severe cognitive, and/or psychiatric impairment, per judgment of NICU and research staff, that precludes cooperation with study protocol
* inability to read, write, speak English or Spanish
* inability or unwillingness to provide signed consent for participation; (5) inability or unwillingness to meet study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Treatment Entry | 8 weeks
  Number of participants having at least one treatment session at a licensed substance use facility or with a licensed counselor
Substance Exposed Pregnancy (SEP) risk as as assessed by a modified Time-Line Follow Back-SEP (TLFB-SEP) | 2 months
  Substance Exposed Pregnancy (SEP) risk as as assessed by a modified Time-Line Follow Back-SEP (TLFB-SEP)
Substance Exposed Pregnancy (SEP) risk as as assessed by a modified Time-Line Follow Back-SEP (TLFB-SEP) | 6 months
  Substance Exposed Pregnancy (SEP) risk as as assessed by a modified Time-Line Follow Back-SEP (TLFB-SEP)
HIV and HCV risk as assessed by Behavioral Risk Assessment for Infectious Disease (BRAID) | 2 months
  HIV and HCV risk as assessed by Behavioral Risk Assessment for Infectious Disease (BRAID)
HIV and HCV risk as assessed by Behavioral Risk Assessment for Infectious Disease (BRAID) | 6 months
  HIV and HCV risk as assessed by Behavioral Risk Assessment for Infectious Disease (BRAID)

SECONDARY OUTCOMES:
Depression as assessed by the Center for Epidemiologic Studies Depression Scale (CES-D) | 2 months
  Depression as assessed by the Center for Epidemiologic Studies Depression Scale (CES-D)
Depression as assessed by the Center for Epidemiologic Studies Depression Scale (CES-D) | 6 months
  Depression as assessed by the Center for Epidemiologic Studies Depression Scale (CES-D)
Current position regarding motivation for change as assessed by the University of Rhode Island Change Assessment (URICA) | 2 months
  Current position regarding motivation for change as assessed by the University of Rhode Island Change Assessment (URICA)
Current position regarding motivation for change as assessed by the University of Rhode Island Change Assessment (URICA) | 6 months
  Current position regarding motivation for change as assessed by the University of Rhode Island Change Assessment (URICA)
Psychological flexibility as assessed by the Acceptance and Action Questionnaire-Substance Abuse (AAQ-SA) | 2 months
  This self-report measure of psychological flexibility will assess a participant's willingness to have undesirable thoughts and feelings related to drug use while still pursuing self-identified goals. This version of the AAQ was specifically developed for substance-abusing populations.
Psychological flexibility as assessed by the Acceptance and Action Questionnaire-Substance Abuse (AAQ-SA) | 6 months
  This self-report measure of psychological flexibility will assess a participant's willingness to have undesirable thoughts and feelings related to drug use while still pursuing self-identified goals. This version of the AAQ was specifically developed for substance-abusing populations.
Number of participants whose infant had routine follow-up pediatric appointments | 6 months
  Medical records will be used, with participant consent, to assess the number of participants whose infant had routine follow-up pediatric appointments.
Number of participants whose infant had acute care visits | 6 months
  Medical records will be used, with participant consent, to assess the number of participants whose infant had acute care visits.
Number of participants whose infant had emergency department visits | 6 months
  Medical records will be used, with participant consent, to assess the number of participants whose infant had emergency department visits.
Number of participants whose infant was re-hospitalized | 6 months
  Medical records will be used, with participant consent, to assess the number of participants whose infant was re-hospitalized.
Number of participants who lost custody of the infant | 6 months
  Medical records will be used, with participant consent, and additionally the research team will collaborate with the NICU social worker and the assigned child protective services (CPS) caseworker, with participant consent, to obtain information about the number of participants who lost custody of the infant.
Number of participants for which any additional abuse or neglect complaints were filed after baseline | 6 months
  Medical records will be used, with participant consent, and additionally the research team will collaborate with the NICU social worker and the assigned child protective services (CPS) caseworker, with participant consent, to obtain information about the number of participants for which any additional abuse or neglect complaints were filed after baseline.
Drug use | 2 months
  Number of participant who test positive for drug use as assessed by urine drug screen
Drug use | 6 months
  Number of participant who test positive for drug use as assessed by urine drug screen

CONTACTS AND LOCATIONS:
Overall Officials: Angela Stotts, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States